CLINICAL TRIAL: NCT03757936
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Recombinant Anti-PD-1 Humanized Monoclonal Antibody Injection (HLX10) in Combination With Recombinant Anti-VEGF Humanized Monoclonal Antibody Injection (HLX04) in Patients With Advanced Solid Tumors
Brief Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Anti-PD-1 Antibody (HLX10) in Combination With Avastin Biosimilar (HLX04) in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10HLX04-001
Record Dates: First submitted 2018-11-19; First posted 2018-11-29 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX04+HLX10 (Experimental): HLX10, at three dose levels (1, 3, 10 mg/kg), to be intravenously injected once every two weeks; HLX04, at a fixed dose of 5 mg/kg, intravenously injected once every two weeks; Study drugs given in combination for up to 2 years or until the disease gets worse, whichever comes first.
  Interventions: Drug: HLX04; Drug: HLX10

INTERVENTIONS:
Drug: HLX04 — Recombinant Anti-VEGF Humanized Monoclonal Antibody Injection
Drug: HLX10 — Recombinant Anti-PD-1 Humanized Monoclonal Antibody Injection

SUMMARY:
This is a single-center, open-label, dose-escalation Phase I clinical trial to evaluate the safety and the tolerability of HLX10-HLX04 combination therapy in patients with advanced solid tumors after failure of standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male or female
2. Patient with histologically or cytologically confirmed advanced malignant solid tumors who have failed standard of care, or has no standard-of-care therapy or are not suitable for standard of care at the present stage;
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1；
4. Life expectancy greater than 3 months;
5. Patient must have at least one measurable tumor lesion as defined by RECIST v1.1; the lesion concerned must not be a bone metastasis if only one target lesion is present;
6. Has adequate organ functions;
7. If the subject is a patient with hepatocellular carcinoma, Child-Pugh classification must be A.
8. A qualified patient (male or female) of childbearing potential must agree to use reliable contraceptive methods (hormonal, or barrier method or abstinence) for the course of the study and through at least 6 months after the last dose; a female patient of childbearing potential must have negative blood pregnancy test within 7 days prior to enrollment;
9. The subject must give his/her informed consent to this study prior to the trial, and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Histopathological confirmed head and neck cancer or squamous-cell lung cancer, or bleeding tendency in the tumor lesion judged by the investigator;
2. Has received antitumor therapy like radiotherapy, chemotherapy, targeted therapy, endocrinal therapy or immunotherapy, or other clinical study drug therapy within 4 months prior to the initial drug administration;
3. Has received a surgical operation on major viscera or experienced apparent trauma within 4 weeks from the initial drug administration, or experienced subcutaneous venous access device implantation within 7 days;
4. The adverse reactions which occurred in the previous antitumor treatment were not recovered to ≤ grade 1 based on CTCAE 4.03 assessment (except for hair loss);
5. Evidences of metastatic lesion in the patient's central nervous system;
6. Previously experienced ≥ grade 3 immune-related adverse event during immunotherapy;
7. Active, or history of autoimmune disease which may relapse (for example, systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.);
8. Currently having or have had interstitial lung disease;
9. Uncontrollable active infection(s);
10. History of immunodeficiency, including HIV antibody positive;
11. Known active hepatitis B; or hepatitis C virus infections;
12. Has bleeding tendency;
13. History of severe cardiovascular diseases;
14. Known gastrointestinal diseases as follows:

    Gastrointestinal perforation, abdominal fistula or abdominal abscess within 6 months before signing the informed consent; History of poorly controlled or recurrent inflammatory bowel disease; Active peptic ulcers, or > moderate esophageal varices;
15. Known hypersensitivity to Bevacizumab, or other anti-PD-1, anti-PD-L1 monoclonal antibody agents;
16. Pregnant or breastfeeding female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-09-27 (Estimated); Study Completion 2020-12-27 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of HLX04 plus HLX10 in patients with advanced solid tumors | 28 days
  The MTD is the dose with toxicity rate (estimated by isotonic regression) most approximate to the target one (30%).
Dose Limiting Toxicity (DLT) of HLX04 plus HLX10 in patients with advanced solid tumors | 28 days
  DLT is defined as the occurrence of the following adverse events (unless judged by the investigator to be definitely unrelated to HLX04 or HLX10) within Cycle 1 (i.e., from Cycle 1 Day 1 to Cycle 1 Day 28)

SECONDARY OUTCOMES:
PK parameters of the HLX04 plus HLX10 therapy in patients with advanced solid tumors | Day 1 of treatment up to 2 years
  Peak Plasma Concentration (Cmax) for single dose and multiple doses
PK parameters of the HLX04 plus HLX10 therapy in patients with advanced solid tumors | Day 1 of treatment up to 2 years
  Area under the plasma concentration versus time curve (AUC) for single dose and multiple doses
Objective Response Rate (ORR) of HLX04 plus HLX10 in patients with advanced solid tumors | Day 1 of treatment up to 2 years
  ORR determined by RECIST criteria
Disease Control Rate (DCR) of HLX04 plus HLX10 in patients with advanced solid tumors | Day 1 of treatment up to 2 years
  DCR determined by RECIST criteria
Duration of Response (DOR) of HLX04 plus HLX10 in patients with advanced solid tumors | Day 1 of treatment up to 2 years
  DOR determined by RECIST criteria
Progression-Free Survival (PFS) of HLX04 plus HLX10 in patients with advanced solid tumors | Day 1 of treatment up to 2 years
  PFS determined by RECIST criteria
Overall Survival (OS) of HLX04 plus HLX10 in patients with advanced solid tumors | Day 1 of treatment up to 2 years
  OS determined by RECIST criteria
Immunogenicity | Day 1 of treatment up to 2 years
  Anti-drug Antibody (ADA) Testing

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No